CLINICAL TRIAL: NCT05129735
Title: An Exploratory Investigation to Assess Changes in Quality of Life for Individuals With Type 2 Diabetes After Taking a Meal-replacement Shake.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrawn
Sponsor: Teatis, Inc (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20227Teatis
Record Dates: First submitted 2021-11-03; First posted 2021-11-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is an open-label single-arm observational trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal replacement shake (Experimental): Teatis meal replacement shake
  Interventions: Dietary Supplement: Meal replacement shake

INTERVENTIONS:
Dietary Supplement: Meal replacement shake — Each day for the study period (12 weeks), the participants will take one meal-replacement shake per day for breakfast. The breakfast will be replaced by the shake entirely.

SUMMARY:
This is an open-label single-arm observational trial to study the effectiveness of a commercially available meal-replacement shake and its effect on the quality of life in individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 18-75 years old
* Diagnosed with type 2 diabetes for at least 3 months
* HbA1c of 7.5 to 10% inclusive
* BMI of 27 to 40 kg/m2
* If on any medication, treated with a stable dose for at least 90 days
* Must be in good health (don't report any medical conditions asked in the screening questionnaire)
* Willing and able to provide written informed consent
* Must have a Glucometer at home

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Have a history of severe hypoglycemia or hyperglycemia requiring hospitalization within the prior 6 months
* Use of dietary supplements or meal-replacement shakes targeted at diabetes and unwilling to stop using them for the duration of the study
* Allergies to any test product ingredients
* Has any of the following medical conditions:
* Oncological conditions
* Psychiatric disease
* Cardiovascular disease: any hospitalization within the past 3 months
* Multiple Sclerosis
* Gastrointestinal conditions such as Celiac disease, Crohn's disease, etc.
* Any other severe chronic disease
* History of drug or alcohol abuse
* Females who are pregnant, want to become pregnant for the duration of the study, or who are breastfeeding during the course of the study
* Participation in a clinical research trial within 30 days prior to screening
* Participating in an investigational health product research study
* Any disorder, unwillingness, or inability, which in the investigator's opinion, might jeopardize the individual's safety or compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of quality of life score from baseline to 12-weeks | 12 weeks
  Survey based quality of life measure on a scale from 0-5 (0=lowest possible score, 5=highest possible score)

SECONDARY OUTCOMES:
Improvement in a1c levels from baseline to 12-weeks | 12 weeks
  Change in a1c biomarkers measured with an at-home blood test after 12 weeks compared to baseline results.
Improvement in blood glucose from baseline to 12-weeks | 12 weeks
  Change in blood glucose biomarkers measured with an at-home blood test after 12 weeks compared to baseline results.
Improvement in insulin levels from baseline to 12-weeks | 12 weeks
  Change in insulin levels measured with an at-home blood test after 12 weeks compared to baseline results.
Improvement in total cholesterol levels from baseline to 12-weeks | 12 weeks
  Change in total cholesterol measured with an at-home blood test after 12 weeks compared to baseline results.
Improvement in triglyceride levels from baseline to 12-weeks | 12 weeks
  Change in triglyceride measured with an at-home blood test after 12 weeks compared to baseline results.
Improvement in HDL cholesterol levels from baseline to 12-weeks | 12 weeks
  Change in HDL cholesterol measured with an at-home blood test after 12 weeks compared to baseline results.
Improvement in LDL cholesterol levels from baseline to 12-weeks | 12 weeks
  Change in LDL cholesterol measured with an at-home blood test after 12 weeks compared to baseline results.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, MSc, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided